CLINICAL TRIAL: NCT07103837
Title: Development, Validity, and Reliability of the Reactive Skill Test in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Ebru Tekin, Pamukkale University, Balikesir University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024/22
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Aging; Cognitive Performance
Keywords: Cognitive-motor testing; Reaction time; Reactive skill

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reactive Skill Test (Experimental)
  Interventions: Other: Reactive Skill Test

INTERVENTIONS:
Other: Reactive Skill Test — The Reactive Skill Test will be conducted using a setup consisting of four pods, white cones, and balls that match the colors of the light signals During the test, a ReactionX device configured with four distinct light colors (red, green, blue, and yellow) will be used. The test protocol is programmed via the ReactionX mobile application to control the sequence and display of lights. Each LED light is illuminated in a randomized order with zero delay time. Upon illumination, the participant is required to select the ball corresponding to the color of the light, place it on the matching cone, and then deactivate the LED light of the same color as the last placed ball. The test concludes once this sequence is completed for all four lights. Performance is evaluated based on parameters such as reaction time, accuracy, and total completion time. This protocol is specifically designed to assess cognitive skills such as color recognition, reaction time, motor coordination, and attention.

SUMMARY:
Aging is associated with cognitive and physical decline, leading to an increased risk of falls in older adults. Recent evidence highlights the critical role of cognitive functions-such as attention, memory, and executive functioning-in postural control and fall risk. This study aims to develop and validate a novel Reactive Skill Test (RST) that simultaneously assesses cognitive (reaction time, visual attention, short-term memory) and motor responses in older adults. The test involves matching colored stimuli to targets using a color-coded pod and cone setup controlled via the ReactionX system. The validity of RST will be examined through correlations with established cognitive and fall risk measures, while test-retest reliability will be assessed across separate sessions. This tool may provide early detection of cognitive-motor impairments contributing to fall risk in aging populations.

ELIGIBILITY:
Inclusion Criteria:

* Being over 60 years of age
* Scoring at least 10 points on the Mini-Mental State Examination (MMSE)
* Ability to ambulate independently
* Being literate
* Providing informed consent to participate in the study

Exclusion Criteria:

* Inability to ambulate independently
* Scoring below 10 points on the Mini-Mental State Examination (MMSE)

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-12-25 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Development of the Reactive Skills Test | For the reliability of RBT, the test will be performed again one week later at the same time of day.
  The Reactive Skill Test will be conducted using a setup consisting of four pods, white cones, and balls that match the colors of the light signals. During the test, a ReactionX device configured with four distinct light colors (red, green, blue, and yellow) will be used. The test protocol is programmed via the ReactionX mobile application to control the sequence and display of lights. Each LED light is illuminated in a randomized order with zero delay time. Upon illumination, the participant is required to select the ball corresponding to the color of the light, place it on the matching cone, and then deactivate the LED light of the same color as the last placed ball. The test concludes once this sequence is completed for all four lights. Performance is evaluated based on parameters such as reaction time, accuracy, and total completion time. This protocol is specifically designed to assess cognitive skills such as color recognition, reaction speed, motor coordination and attention.

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) | the first day of inclusion in the study, once
  The Mini-Mental State Examination (MMSE) is widely recognized as one of the most commonly used tools for assessing cognitive impairment worldwide. The MMSE evaluates orientation, memory, attention, calculation, recall, language, motor function, perception, and visuospatial abilities. Its ease and rapid administration are among its main advantages. In this study, the MMSE will be used to assess cognitive function. Scores ranging from 27 to 30 are considered normal, 24 to 27 indicate mild cognitive impairment, 20 to 23 represent mild dementia, 10 to 19 correspond to moderate dementia, and scores below 10 indicate severe dementia.
Five Times Sit-to-Stand Test (FTSST) | the first day of inclusion in the study, once
  The Five Times Sit-to-Stand Test is a standardized assessment used to evaluate lower extremity muscle strength and balance in older adults. Participants sit on a backless chair 45 cm in height with their arms crossed over their chest and are instructed to stand up and sit down five times as quickly as possible. Performance is measured by timing the duration from the initial seated position to the final seated position using a stopwatch. The validity of the test is supported by its correlation with measures of knee extension strength and walking performance. It assesses lower limb strength and functional mobility. Times exceeding 15 seconds are associated with a higher risk of falls. The test will be performed three times, and the average time will be recorded.
International Physical Activity Questionnaire (Short Form) | the first day of inclusion in the study, once
  This questionnaire will be used to assess participants' physical activity levels in daily life. Participants report the types of activities performed and the time spent on each over the past seven days. Walking, sitting, moderate-intensity, and vigorous-intensity activities will be recorded based on participant self-report. The score is calculated by multiplying the MET value assigned to each activity by the duration and the number of days performed per week, resulting in a MET-minutes/week value. MET values are assigned as follows: walking = 3.3 MET, moderate activity = 4 MET, and vigorous activity = 8 MET. Based on these scores, participants will be classified into three categories: physically inactive (<600 MET-min/week), low physical activity level (600-1500 MET-min/week), and sufficient physical activity level (>1500 MET-min/week).
Hand Reaction Time Test | the first day of inclusion in the study, once
  Hand movement reaction times will be recorded using an LED light system connected to a smartphone application (ReactionX). The ReactionX system consists of six LEDs and a wireless lighting setup. Participants will be seated with both hands placed on the table, palms down, spaced 40 cm apart (ReactionX device positioned centrally, 20 cm from each hand) and elbows flexed at 90°. When a light illuminates, participants are instructed to touch the device with the indicated hand as quickly as possible to turn off the light. Each test will be performed six times, with the best trial recorded. Results will be expressed in milliseconds (ms).

CONTACTS AND LOCATIONS:
Locations (1):
- Balikesir University, Balıkesir, Bigadiç, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No